CLINICAL TRIAL: NCT03905928
Title: Establishing the Effect of Flavor on the Addictive Potential of Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andrea Hobkirk, PhD, Assitant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 11837; R03DA047582 (NIH)
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Dependence
Keywords: smoking; electronic cigarettes; flavor; cue-reactivity
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Vaping

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 18mg/ml Tobacco Flavor ECIG (Experimental): Participants will be provided with an ECIG containing 18mg/ml nicotine concentration and a tobacco flavor.
  Interventions: Other: Nicotine Containing ECIG with tobacco flavor
- 0mg/ml Tobacco Flavor ECIG (Placebo Comparator): Participants will be provided with an ECIG containing 0mg/ml nicotine concentration and a tobacco flavor.
  Interventions: Other: Placebo ECIG with Tobacco Flavor
- 18mg/ml Strawberry Vanilla Flavor ECIG (Experimental): Participants will be provided with an ECIG containing 18mg/ml nicotine concentration and a strawberry vanilla flavor.
  Interventions: Other: Nicotine Containing ECIG with Strawberry Vanilla Flavor
- 0mg/ml Strawberry Vanilla Flavor ECIG (Placebo Comparator): Participants will be provided with an ECIG containing 0mg/ml nicotine concentration and a strawberry vanilla flavor.
  Interventions: Other: Placebo ECIG with Strawberry Vanilla Flavor

INTERVENTIONS:
Other: Nicotine Containing ECIG with tobacco flavor — Participants will be provided with an EGO style ECIG to be used for 28 days. The EGO style ECIG is a "vape pen-style" device that comprises of a rechargeable battery and a tank containing liquid. Those in this intervention group will receive an ECIG with 18mg/ml nicotine concentration and a tobacco flavor.
  Arms: 18mg/ml Tobacco Flavor ECIG
Other: Nicotine Containing ECIG with Strawberry Vanilla Flavor — Participants will be provided with an EGO style ECIG to be used for 28 days. The EGO style ECIG is a "vape pen-style" device that comprises of a rechargeable battery and a tank containing liquid. Those in this intervention group will receive an ECIG with 18mg/ml nicotine concentration and a strawberry vanilla flavor.
  Arms: 18mg/ml Strawberry Vanilla Flavor ECIG
Other: Placebo ECIG with Tobacco Flavor — Participants will be provided with an EGO style ECIG to be used for 28 days. The EGO style ECIG is a "vape pen-style" device that comprises of a rechargeable battery and a tank containing liquid. Those in this intervention group will receive an ECIG with 0mg/ml nicotine concentration and a tobacco flavor.
  Arms: 0mg/ml Tobacco Flavor ECIG
Other: Placebo ECIG with Strawberry Vanilla Flavor — Participants will be provided with an EGO style ECIG to be used for 28 days. The EGO style ECIG is a "vape pen-style" device that comprises of a rechargeable battery and a tank containing liquid. Those in this intervention group will receive an ECIG with 0mg/ml nicotine concentration and a strawberry vanilla flavor.
  Arms: 0mg/ml Strawberry Vanilla Flavor ECIG

SUMMARY:
The current study aims to establish proof-of-concept that neural cue-reactivity can serve as an early, objective marker of electronic cigarette (ECIG) addictive potential. Further, this study will examine the effect of flavor and nicotine concentration on the addictive potential of ECIGs to aid research informing U.S. Food and Drug Administration (FDA) flavor regulations and smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21-60
2. Smoke filtered cigarettes/machine-rolled cigarettes (≥5 cigarettes per day) or daily e-cigarette use for past year.
3. No serious quit attempt in prior month. This includes use of any FDA approved smoking cessation medication (varenicline, bupropion [used specifically as a quitting aid], patch, gum, lozenge, inhaler, and nasal spray) in the past 1 month as an indication of treatment seeking.
4. Willing to supplement cigarette smoking with ECIG use for 4 weeks or replace e-cigarette with study product for 4 weeks
5. Willing to attend regular visits over a 4-week period (not planning to move, not planning extended vacation, no planned surgeries)
6. Willing to undergo two fMRI scans
7. Able to read and write in English
8. Able to understand and consent to study procedures
9. Access to computer with internet service that allows for use of Zoom

Exclusion Criteria:

1. Impaired smell function as measured via a standardized screening assessment
2. Unstable or significant medical condition in the past 12 months (recent heart attack or some other heart conditions, stroke, severe angina including high blood pressure)
3. Severe immune system disorders (uncontrolled Human Immunodeficiency virus infection; unstable multiple sclerosis symptoms), respiratory diseases (exacerbations of asthma or chronic obstructive pulmonary disorder, require oxygen, require oral prednisone), kidney (dialysis) or liver diseases (cirrhosis), or any medical disorder/medication that may affect participant safety or biomarker data
4. Women who are pregnant (verified by urine pregnancy test at any visit), trying to become pregnant, or nursing
5. Medical conditions associated with cognitive impairment or neurological dysfunction
6. Severe claustrophobia
7. Current depressive or anxiety disorder
8. Uncontrolled mental illness or substance abuse or inpatient treatment for these conditions in the past 6 months
9. Use of illicit drugs or prescription drugs for non-medical use daily/almost daily or weekly in the past 3 months per National Institute on Drug Abuse (NIDA) Quick Screen, not including use of marijuana
10. Any known risk from exposure to high-field strength magnetic fields (e.g., cardiac pacemakers), any irremovable metallic foreign objects in their body (e.g., braces), or a questionable history of metallic fragments which are likely to create artifact on the MRI scans
11. Known allergy to propylene glycol or vegetable glycerin
12. Other member of household currently participating in the study
13. History of a seizure disorder or had a seizure in the past 12 months
14. Currently taking medications prescribed to prevent seizures (such as Carbamazepine or Phenobarbital). Using seizure medications for off-label use (indications other than treatment for seizures) will not be included as an exclusion, these will be assessed on a case-by-case basis

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 18mg/ml Tobacco Flavor ECIG | 0mg/ml Tobacco Flavor ECIG | 18mg/ml Strawberry Vanilla Flavor ECIG | 0mg/ml Strawberry Vanilla Flavor ECIG
Started | 6 | 3 | 5 | 5
Completed | 5 | 3 | 3 | 4
Not Completed | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18mg/ml Tobacco Flavor ECIG | 0mg/ml Tobacco Flavor ECIG | 18mg/ml Strawberry Vanilla Flavor ECIG | 0mg/ml Strawberry Vanilla Flavor ECIG | Total
Number analyzed (Participants) | 6 | 3 | 5 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.00 (9.30) | 41.67 (13.05) | 45.60 (10.46) | 44.40 (8.99) | 46.00 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 4 | 13
  Male | 2 | 1 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 3 | 4 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 2 | 5 | 5 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline Neural Flavor Cue-reactivity at Baseline
Description: Functional magnetic resonance imaging (fMRI) will be used to measure blood oxygen-level dependent (BOLD) signal in response to tobacco vs. strawberry-vanilla ECIG flavors at baseline. The means reported are the average percentage of BOLD signal change between the fMRI task odor conditions (tobacco vs. strawberry) identified using a whole-brain one-sample t-test with FSL software. Positive values indicate stronger BOLD signal during tobacco odor cues and negative values indicate stronger BOLD signal during strawberry odor cues.
Time Frame: Baseline
Population: For this within-subjects comparison of laboratory task conditions, we included all 19 participants who completed a functional MRI scan at baseline. All assigned groups were combined since group assignment was not a variable of interest for this aim.
Measure: Mean (Standard Deviation); unit: percentage of BOLD signal change
Groups:
- Total Baseline Sample: The total baseline sample includes the 19 participants who completed a functional MRI scan at baseline and were randomized to a condition, regardless of study completion.
Arm/Group | Total Baseline Sample
Number analyzed (Participants) | 19
percentage of BOLD signal change
  Right insula | 0.08 (0.07)
  Left amygdala | 0.23 (0.20)
  Ventral tegmental area | 0.10 (0.07)
  Left ventral cerebellum | 0.14 (0.12)
  Right dorsal cerebellum | 0.13 (0.16)
  Left dorsal cerebellum | 0.09 (0.07)
  Medial prefrontal cortex | -0.15 (0.13)
  Left medial pre/postcentral gyri | -0.06 (0.05)
  Left lateral pre/postcentral gyri | -0.07 (0.07)
  Precuneous | -0.07 (0.06)
  Right pre/postcentral gyri | -0.06 (0.04)
  Bilateral superior frontal gyrus | -0.07 (0.05)
Statistical Analysis 1: Comparison: Total Baseline Sample; This was a whole-brain, voxel-wise general linear model conducted in FSL software using a one-sample t-test on the tobacco>strawberry condition contrasts conducted at the subject-level; Test type: Superiority; A whole-brain, one-sample t-test was used with a voxel threshold p <.001 and cluster threshold p<.05. This method results in unique p-values for each cluster identified

2. Primary Outcome: Changes in Neural Flavor Cue-reactivity Across Nicotine Groups
Description: Functional magnetic resonance imaging (fMRI) will be used to measure changes in blood oxygen-level dependent (BOLD) signal for the tobacco>strawberry contrast across 18 mg/ml vs. 0 mg/ml nicotine concentration groups from baseline to 4-weeks post-randomization using a whole-brain repeated measures ANOVA with FSL software. The means reported are the difference (4-week post-intervention - baseline) of the average percentage of BOLD signal change between the fMRI task odor conditions (tobacco vs. strawberry). Positive values indicate increases in tobacco>strawberry BOLD signal and negative values indicate decreases in tobacco> strawberry BOLD signal.
Time Frame: Baseline to 4-weeks
Population: This analysis includes 15 participants who completed baseline and post-intervention functional MRI scans. Groups assigned to nicotine vs. no nicotine were compared and flavor sub-groups within the nicotine groups (tobacco vs. strawberry) were combined, since flavor was not a variable of interest for this aim.
Measure: Mean (Standard Deviation); unit: % BOLD signal change difference score
Groups:
- 18 mg/ml Nicotine Concentration E-cigarettes: This group includes participants randomized to the 18 mg/ml nicotine concentration e-cigarettes, regardless of flavor.
- 0 mg/ml Nicotine Concentration E-cigarettes: This group includes participants randomized to the 0 mg/ml nicotine concentration e-cigarettes, regardless of flavor.
Arm/Group | 18 mg/ml Nicotine Concentration E-cigarettes | 0 mg/ml Nicotine Concentration E-cigarettes
Number analyzed (Participants) | 8 | 7
% BOLD signal change difference score
  Left insula | 0.18 (0.17) | -0.12 (0.15)
  Medial prefrontal cortex | 0.21 (0.14) | -0.21 (0.29)
Statistical Analysis 1: Comparison: 18 mg/ml Nicotine Concentration E-cigarettes vs 0 mg/ml Nicotine Concentration E-cigarettes; This was a whole-brain, voxel-wise repeated measures ANOVA conducted using FSL software on activation from baseline to post-intervention that differ by the nicotine groups (18 mg/ml vs. 0 mg/ml) for the tobacco>strawberry condition contrasts calculated at the subject-level. The means and standard deviations presented are the average post-pre scan difference scores of the BOLD percentage signal change of tobacco > strawberry contrasts for each group; Test type: Superiority; A whole-brain, repeated measures ANOVA was used with a voxel threshold p <.025 and cluster threshold p<.05. This method results in unique p-values for each cluster identified

3. Primary Outcome: Changes in Neural Flavor Cue-reactivity Across Flavor Groups
Description: Functional magnetic resonance imaging (fMRI) will be used to measure changes in blood oxygen-level dependent (BOLD) signal for the tobacco > strawberry contrast across flavor groups (tobacco vs. strawberry) from baseline to 4-weeks post-randomization. The means reported are the difference (4-week post-intervention - baseline) of the average percentage of BOLD signal change between the fMRI task odor condition (tobacco vs. strawberry) identified using a whole-brain repeated measures ANOVA with FSL software. Positive values indicate increases in tobacco>strawberry BOLD signal and negative values indicate decreases in tobacco> strawberry BOLD signal.
Time Frame: Baseline to 4-weeks
Population: This analysis includes 15 participants who completed baseline and post-intervention functional MRI scans. Groups assigned to tobacco vs. strawberry were compared and nicotine sub-groups within the flavor groups (nicotine vs. no nicotine) were combined, since nicotine was not a variable of interest for this aim.
Measure: Mean (Standard Deviation); unit: % BOLD signal change difference score
Groups:
- Tobacco Flavor: Participants randomized to use an e-cigarette with tobacco-flavored e-liquid, regardless of nicotine concentration.
- Strawberry Flavor: Participants randomized to use an e-cigarette with strawberry-vanilla flavored e-liquid, regardless of nicotine concentration.
Arm/Group | Tobacco Flavor | Strawberry Flavor
Number analyzed (Participants) | 8 | 7
% BOLD signal change difference score
  Right prefrontal cortex | -0.07 (0.03) | 0.05 (0.05)
  Thalamus and right insula | -0.05 (0.01) | 0.06 (0.06)
Statistical Analysis 1: Comparison: Tobacco Flavor vs Strawberry Flavor; This was a whole-brain, voxel-wise repeated measures ANOVA conducted using FSL software on activation from baseline to post-intervention between the flavor groups (tobacco vs. strawberry) for the tobacco>strawberry condition contrasts calculated at the subject-level. The means and standard deviations presented are the average post-pre scan difference scores of the BOLD percentage signal change of tobacco > strawberry contrasts for each group; Test type: Superiority; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: ECIG Dependence
Description: Changes in self-reported ECIG dependence will be measured using the Penn State Electronic Cigarette Dependence Index (PSECDI). Total scores on this 10-item measure range from 0 to 20, with higher scores indicating higher levels of e-cigarette dependence. The means reported here are the week 4 - week 2 difference scores of the total dependence score. Positive means indicate increases in e-cigarette dependence, while negative means indicated decreases in e-cigarette dependence.
Time Frame: 2-weeks post-randomization to 4-weeks post-randomization
Population: This analysis included 14 participants who completed the 2-week check-in and 4-week post-intervention visits and completed the PSECDI.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 18mg/ml Tobacco Flavor ECIG: Participants will be provided with an ECIG containing 15mg/ml nicotine concentration and a tobacco flavor.
- 18mg/ml Strawberry Vanilla Flavor ECIG: Participants will be provided with an ECIG containing 15mg/ml nicotine concentration and a strawberry vanilla flavor.
Arm/Group | 18mg/ml Tobacco Flavor ECIG | 0mg/ml Tobacco Flavor ECIG | 18mg/ml Strawberry Vanilla Flavor ECIG | 0mg/ml Strawberry Vanilla Flavor ECIG
Number analyzed (Participants) | 5 | 3 | 2 | 4
units on a scale | -1.60 (2.07) | -1.33 (3.21) | -3.00 (4.24) | 0.00 (1.41)
Statistical Analysis 1: Comparison: 18mg/ml Tobacco Flavor ECIG vs 0mg/ml Tobacco Flavor ECIG vs 18mg/ml Strawberry Vanilla Flavor ECIG vs 0mg/ml Strawberry Vanilla Flavor ECIG; We conducted a one-way ANOVA to compare the change in e-cigarette dependence (week 4 - week 2 PSECDI difference score) between the four e-cigarette groups; Test type: Superiority; p = 0.573, ANOVA

5. Secondary Outcome: ECIG Liking and Satisfaction
Description: Changes in subjective experiences of ECIG use related to liking and satisfaction will be collected via a self-report survey. The survey consists of 21-items (7-reversed scored) with response options on a 7-point likert scale and total scores ranging from 0 to 126. Higher scores indicate more ECIG liking and satisfaction. The means reported here are the difference of the total scores at week 4 - week 2, with positive means indicating increases in e-cigarette liking and negative means indicating decreases in liking. Note that standard deviation cannot be reported for groups with only one participant.
Time Frame: 2-weeks to 4-weeks
Population: This analysis includes 8 participants who completed the e-cigarette evaluation scale at the 2-week check-in and 4-week post-intervention visit. Only participants who reported using the study e-cigarette since the last study visit completed the evaluation scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 18mg/ml Tobacco Flavor ECIG | 0mg/ml Tobacco Flavor ECIG | 18mg/ml Strawberry Vanilla Flavor ECIG | 0mg/ml Strawberry Vanilla Flavor ECIG
Number analyzed (Participants) | 3 | 1 | 1 | 3
units on a scale | 2.33 (7.57) | -21.00 (0.00) | 16 (0.00) | -5.00 (4.36)

6. Secondary Outcome: Craving to Smoke/Vape
Description: Changes in self-reported craving to smoke/vape were measured with 3 questions on amount, intensity, and self-control using visual analogue scales ranging from 0 to 10 prior to completing the functional MRI scan. Total scores range from 0 to 30 and higher scores indicate more craving. The means reported here are week 4 post-intervention - baseline difference scores of the total craving score. Positive means indicate increases in craving, while negative means indicate decreases in craving.
Time Frame: Baseline to 4-weeks post-randomization
Population: This analysis includes 15 participants that completed the craving scales before the functional MRI scans at baseline and at the post-intervention visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 18mg/ml Tobacco Flavor ECIG | 0mg/ml Tobacco Flavor ECIG | 18mg/ml Strawberry Vanilla Flavor ECIG | 0mg/ml Strawberry Vanilla Flavor ECIG
Number analyzed (Participants) | 5 | 3 | 3 | 4
units on a scale | 3.00 (5.43) | 3.00 (5.43) | -11.00 (2.65) | 1.50 (4.43)
Statistical Analysis 1: Comparison: 18mg/ml Tobacco Flavor ECIG vs 0mg/ml Tobacco Flavor ECIG vs 18mg/ml Strawberry Vanilla Flavor ECIG vs 0mg/ml Strawberry Vanilla Flavor ECIG; We conducted a one-way ANOVA to compare changes in self-reported craving across all groups; Test type: Superiority; p = .022, ANOVA

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | 18mg/ml Tobacco Flavor ECIG | 0mg/ml Tobacco Flavor ECIG | 18mg/ml Strawberry Vanilla Flavor ECIG | 0mg/ml Strawberry Vanilla Flavor ECIG
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 1/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18mg/ml Tobacco Flavor ECIG (N=6) | 0mg/ml Tobacco Flavor ECIG (N=3) | 18mg/ml Strawberry Vanilla Flavor ECIG (N=5) | 0mg/ml Strawberry Vanilla Flavor ECIG (N=5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant experienced mild throat irritation during the first few days of using the e-cigarette.
Procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant had fluid drained from knee after experiencing pain.
Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant experienced flu-like symptoms they reported were related to seasonal allergies.

LIMITATIONS AND CAVEATS:
Results of brain activation reported here are average values of the percentage of blood-oxygen level-dependent signal change (tobacco vs. strawberry task odor conditions) extracted after conducting whole-brain, voxel-wise general linear models with FSL software. The sample size was too small to conduct some planned between-group analyses and significance thresholds were increased for some analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03905928/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03905928/ICF_001.pdf